CLINICAL TRIAL: NCT03140046
Title: Visual Outcomes of Topography Guided Photorefractive Keratectomy (PRK) for Treatment of Patients With Irregular Cornea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelsamee Mohammed, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRK
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Irregular Astigmatism
MeSH Terms: interventions — Photorefractive Keratectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corneal Topography (Experimental): we will do Corneal Topography for every patient before doing photorefractive keratectomy (PRK) and also after it , to measure the change in the quality of vision and measure the change in the quality of vision
  Interventions: Procedure: photorefractive keratectomy (PRK)

INTERVENTIONS:
Procedure: photorefractive keratectomy (PRK) — The cornea will be ablated while the patient fixating on target light under constant eye-tracking control. The ablations will be made using the "ALLEGRETTO X 500WAVE excimer laser" (WaveLight Laser Technologie AG).
  Other Names: PRK

SUMMARY:
Irregular astigmatism is one of the most serious and frequent complications of corneal refractive surgery and one of the worst sequelae of other forms of corneal surgery . It is also considered as one of common, serious complications of corneal injuries .

Spectacle correction is usually not useful in the correction of corneal irregular astigmatism. Contact lenses represent a good alternative, but their adaptation and stability are limited by the irregular corneal surface and patient discomfort.

In recent years, advancements in laser technology have offered better tools for dealing with irregular astigmatism with finding new surgical methods to improve corneal regularity for the correction of irregular astigmatism.

Topography-linked excimer laser is a potentially effective technique in the treatment of irregular astigmatism after keratoplasty . In fact, customized ablation was shown to be an effective means of treatment of irregular astigmatism due to different etiologies Such as corneal Injuries , scar , or postoperative.

Some of the theoretical advantages of topography-driven photorefractive keratectomy (PRK) are a better astigmatic correction, the possibility of correcting irregular astigmatism, and a smaller ablation volume compared with standard treatments, resulting in better visual performance.

Aim of the work To evaluate the efficacy, safety, and predictability of topography-guided photorefractive keratectomy (PRK) to improve refractive status of patient with irregular Cornea.

ELIGIBILITY:
Inclusion Criteria:

* Patients with irregular corneal astigmatism caused by:

  * Trauma.
  * Non - Central Corneal Scars.
  * Previous corneal surgery.
* With No other abnormalities in the eye.
* Patient is willing to enter the study and sign a consent.

Exclusion Criteria:

* Patients with central corneal scars.
* Patients with central haze interfering with visual acuity.
* Patients with ectasia at corneal graft margins.
* Patients with irregular astigmatism caused by corneal ectasia or keratoconus.
* Patients had refractive surgery with ablations leaving a residual corneal thickness less than 250 μm.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | follow up after 1 day, 1 week, 1 month and 3 months
  The measure of the Visual Acuity and Best Corrected Visual acuity Using the Snellen Chart which give use an idea about visual acuity in Metric scale (e.g. 6\6 , 6\12)

SECONDARY OUTCOMES:
Refractive State | follow up after 1 day, 1 week, 1 month and 3 months
  We will measure the Refractive state of the eye by using the Auto refractor which give us an idea about the refractive state in a Diopteric scale ( e.g. -2D , +4 D) .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No